CLINICAL TRIAL: NCT00003147
Title: Phase I Study of Percutaneous Injections of Adeno-Virus p53 Construct (ADENO-p53) for Hepatocellular Carcinoma
Brief Title: Gene Therapy in Treating Patients With Cancer of The Liver
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02259; PCI-96-035; NCI-T96-0059; CDR0000065932 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-04-06; First posted 2004-08-24 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2000-05

CONDITIONS: Liver Cancer
Keywords: localized unresectable adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — advexin

ARMS (1):
- Arm I (Experimental): Patients receive adenovirus p53 construct by percutaneous injection to a maximum of two lesions on day 1. Treatment is repeated every 28 days for up to 6 courses. In the absence of dose-limiting toxicity (DLT) in the first cohort of 6 patients treated, subsequent cohorts of 6 patients each receive escalating doses of the drug on the same schedule. If DLT occurs in 2 of 6 patients at a given dose level, then dose escalation ceases and that dose is declared the maximum tolerated dose. Study treatment may continue in the absence of disease progression and unacceptable adverse events.
  Interventions: Biological: Ad5CMV-p53 gene

INTERVENTIONS:
Biological: Ad5CMV-p53 gene

SUMMARY:
Phase I trial to study the effectiveness of gene therapy with the p53 gene in treating patients who have cancer of the liver that cannot be surgically removed. Inserting the p53 gene into a person's tumor may improve the body's ability to fight liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the safety of adenovirus p53 construct (adeno-p53) in patients with hepatocellular carcinoma.

II. Investigate the potential effects of intralesional adeno-p53 given by monthly percutaneous injections in these patients.

OUTLINE: This is a dose escalation, multicenter study.

Patients receive adenovirus p53 construct by percutaneous injection to a maximum of two lesions on day 1. Treatment is repeated every 28 days for up to 6 courses. In the absence of dose-limiting toxicity (DLT) in the first cohort of 6 patients treated, subsequent cohorts of 6 patients each receive escalating doses of the drug on the same schedule. If DLT occurs in 2 of 6 patients at a given dose level, then dose escalation ceases and that dose is declared the maximum tolerated dose. Study treatment may continue in the absence of disease progression and unacceptable adverse events.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed unresectable hepatocellular carcinoma (HCC) or highly suspicious for HCC based on CT scan and elevated alfafetoprotein
* Measurable disease by abdominal CT scan Accessible (peripheral) lesions
* No metastatic disease

PATIENT CHARACTERISTICS:

* Age: Over 18
* Performance status: ECOG 0-2
* Life expectancy: At least 12 weeks
* Platelet count at least 60,000/mm3
* Absolute neutrophil count greater than 1,500/mm3
* Prothrombin time of no greater than 16 seconds after administration of fresh frozen plasma
* Bilirubin no greater than 3.0 mg/dL
* Creatinine less than 1.5 mg/dL
* Child's class A or B cirrhosis eligible
* No uncontrolled infection Not pregnant or breast feeding
* No unstable or severe intercurrent medical condition

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior chemotherapy
* At least 4 weeks since prior radiation therapy
* No prior hepatic transplantation
* No more than 1 prior systemic regimen for hepatocellular carcinoma allowed
* No concurrent therapy with other investigational agents
* No prior gene therapy
* No prior intralesional therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1998-02; Primary Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandra P. Belani, MD, Study Chair — University of Pittsburgh
Locations (2):
- United States (2):
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania